CLINICAL TRIAL: NCT00816621
Title: Early Intervention for Children Adopted Internationally
Brief Title: Effectiveness of a Parent Training Program for Parents of Children Adopted Internationally
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Delaware (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Mary Dozier, Principal Investigator, University of Delaware
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: R01MH084135 (NIH); R01MH084135 (NIH); DSIR 84-CTP
Record Dates: First submitted 2008-12-30; First posted 2009-01-01 (Estimated); Last update posted 2021-06-02 (Actual); Status verified 2021-05

CONDITIONS: Attachment Disorders
Keywords: Internationally Adopted Children; Adoption; Attachment; Inattention; Prevention
MeSH Terms: interventions — abacavir; butyl phosphorotrithioate; Physical Therapy Modalities; Occupational Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ABC for Children Adopted Internationally (Experimental): ABC for Children Adopted Internationally: 10 session in home intervention that targets parent nurturance, synchrony, pseudo-autistic behaviors, and indiscriminate sociability
  Interventions: Behavioral: ABC for Children Adopted Internationally
- DEF for Children Adopted Internationally (Active Comparator): DEF for Children Adopted Internationally: 10 session in home intervention that targets cognitive and motor delays
  Interventions: Behavioral: DEF for Children Adopted Internationally

INTERVENTIONS:
Behavioral: ABC for Children Adopted Internationally — Participants will participate in 10 weekly in-home intervention sessions aimed at enhancing the ability of children to regulate their attention, behavior, and physiology and to develop secure, organized attachments to their parents.
  Other Names: Attachment and Biobehavioral Catch-up; ABC; ABC-I
  Arms: ABC for Children Adopted Internationally
Behavioral: DEF for Children Adopted Internationally — Participants will participate in 10 weekly in-home intervention sessions aimed at enhancing the intellectual and language development of children.
  Other Names: DEF; PT/OT; Physical Therapy/Occupational Therapy
  Arms: DEF for Children Adopted Internationally

SUMMARY:
This study will test the effectiveness of a parent training program aimed at helping children who are adopted internationally to develop secure, organized attachments to their parents.

DETAILED DESCRIPTION:
Children adopted internationally by parents in the United States often experience institutional care prior to adoption. Early institutional care may lead to inattention, deficits in inhibitory control, and insecure attachments in children. Many of these problems persist even after the child is adopted. This study will test the effectiveness of a parent training program called Attachment and Biobehavioral Catch-up for Children Adopted Internationally (ABC-I). This program is designed to enhance children's ability to regulate their attention, behavior, and physiology and to develop secure, organized attachments to their parents.

Participation in this study will begin when the child participant is between 12 and 20 months old, and it will end when the child is 4 years old. Participants, who will include parents and their adopted child, will meet with the study researchers 3 times before receiving the training program intervention, twice in their home and once at the research site. During these visits, the background and medical history of the child participant will be reviewed. Participants will then be randomly assigned to receive 1 of 2 parent training programs: ABC-I or Developmental Education for Families (DEF). Both programs will involve 10 weekly sessions, each lasting 60 to 90 minutes and occurring in the parents' homes. The DEF training program will focus on enhancing the intellectual and language development of the child participant, but it will not train parents to pay attention to and interpret their children's cues. The ABC-I training program will involve videotaping parents while they interact with their children, reviewing the videotapes, discussing strategies for interacting with children, and completing homework assignments.

Participants will undergo assessments before and after the training programs and at follow-up visits when each child turns 2, 3, and 4 years old. Assessments will be made of sensitivity in parents and of inattention, inhibitory control, attachment quality, and cortisol production in children. Parent sensitivity will be measured by observing parent-child interactions and coding them according to a pre-existing scale. Child inattention and inhibitory control will be measured through observing each child's behaviors on various structured tasks, such as watching a video with a distracter present or being told to wait to open a wrapped gift. Attachment will be measured through observation of child behavior and through parent ratings and diaries. Cortisol production will be measured through a saliva sample, collected via cotton swab. When children are 4 years old, they will also be evaluated for diagnosable behavioral disorders. For a subset of children, cheek swabs will be collected at age 5-6 for the assessment of telomere length.

ELIGIBILITY:
Inclusion Criteria:

* Adopted a child internationally

Exclusion Criteria:

* Child has known serious medical condition, such as cerebral palsy

Ages: 12 Months to 36 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2009-01 (Actual); Primary Completion 2020-12-10 (Actual); Study Completion 2021-03-20 (Actual)

PRIMARY OUTCOMES:
Inattention | Measured pre-intervention, post-intervention, and when the child turns 2, 3, and 4

SECONDARY OUTCOMES:
Cortisol production | Measured pre-intervention, post-intervention, and when the child turns 2, 3, and 4
  Salivary cortisol measured at wake-up and bedtime. Eliza assay will be used.
Competence | Measured post-intervention at ages 3 and 4
  Observational protocol from Disruptive Behaviors-Diagnostic Observation Scale (DB-DOS)
Problem behaviors | Measured post-intervention at ages 3 and 4
  Observational protocol (DB-DOS)
Attachment | Measured post-intervention at age 2-4
  "Strange Situation" - lab based assessment
Executive functioning | Measured at ages 3 and 4
  Dimensional change card sort
Emotion regulation | Measured at ages 3 and 4
  Perfect circle
Problem behaviors | Ages 3 and 4
  Child Behavior Checklist
Executive functioning | Ages 3 and 4
  Day-night Stroop

CONTACTS AND LOCATIONS:
Overall Officials: Mary Dozier, PhD, Principal Investigator — University of Delaware
Locations (1):
- University of Delaware, Newark, Delaware, United States

REFERENCES:
- [Derived] Yarger HA, Lind T, Raby KL, Zajac L, Wallin A, Dozier M. Intervening With Attachment and Biobehavioral Catch-Up to Reduce Behavior Problems Among Children Adopted Internationally: Evidence From a Randomized Controlled Trial. Child Maltreat. 2022 Aug;27(3):478-489. doi: 10.1177/10775595211010975. Epub 2021 Apr 22. PMID 33882710
- [Derived] Lind T, Lee Raby K, Goldstein A, Bernard K, Caron EB, Yarger HA, Wallin A, Dozier M. Improving social-emotional competence in internationally adopted children with the Attachment and Biobehavioral Catch-up intervention. Dev Psychopathol. 2021 Aug;33(3):957-969. doi: 10.1017/S0954579420000255. PMID 32672145
- [Derived] Yarger HA, Bernard K, Caron EB, Wallin A, Dozier M. Enhancing Parenting Quality for Young Children Adopted Internationally: Results of a Randomized Controlled Trial. J Clin Child Adolesc Psychol. 2020 May-Jun;49(3):378-390. doi: 10.1080/15374416.2018.1547972. Epub 2019 Jan 16. PMID 30649970